CLINICAL TRIAL: NCT04896190
Title: The Relationship Between Q Angle and Quadriceps Muscle Activation on Dynamic Balance in Women
Acronym: Quadriceps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, merve yilmaz menek, Principle investigator, Istanbul Medipol University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: merveyilmaz
Record Dates: First submitted 2021-05-13; First posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Physiotherapy and Rehabilitation
Keywords: Q angle; Quadriceps muscle activation; EMG; Balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Before the evaluation of EMG amplitude on dynamic balance position, the Q angle was measured in supine and standing positions. The EMG signals collected by measuring the muscle activation of the Vastus Medialis and Vastus Lateralis during dynamic balance position on the ProKin device were recorded. Q angle evaluations, static and dynamic balance and functional status of all participants were evaluated.
  Interventions: Other: Evaluation of Q angle and Quadriceps muscle activation on dynamic balance position

INTERVENTIONS:
Other: Evaluation of Q angle and Quadriceps muscle activation on dynamic balance position — Evaluation of Q angle, Quadriceps muscle activation, static and dynamic balance and functionality of all individuals was done.

SUMMARY:
The quadriceps angle (Q angle) is significant for the lower extremity alignment. Anatomical alignment of Q angle is related to Quadriceps muscle strength. Women have consistently been found to have larger Q angles than men and are more often affected due to patellofemoral problems. Quadriceps muscle activation and lower extremity alignment affect musculoskeletal health in women.The aim of this study wa s to determine the relationship between Q angle and quadriceps muscle activation on dynamic balance in women.

DETAILED DESCRIPTION:
Objective: To determine the relationship between Q angle and quadriceps muscle activation on dynamic balance in women. Design: Correlational Study. Setting: University. Participants: Forth women will be included in the study. Interventions: Q angle in standing and supine positions, quadriceps muscle activation, static and dynamic balance and functionality were measured. Main Outcome Measurements: Q angle will measured with a tape measure; muscle activation will measured with Surface Electromyography (EMG) static balance will measured with Flamingo Balance Test (FBT); dynamic balance will measured with ProKin 252 Techno Body device; and, functionality will measured with Short Form Musculoskeletal Assessment (SFMA). Before the evaluation of EMG amplitude on dynamic balance position, the Q angle will measured in supine and standing positions. The EMG signals collected by measuring the muscle activation of the Vastus Medialis and Vastus Lateralis during dynamic balance position on the ProKin device will recorded.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were being women, being aged 19-25, and not having musculoskeletal or neurological problems.

Exclusion Criteria:

* Exclusion criteria were having an operation in the past year, taking medicine related to lower limb problems, persistent pain and discomfort of the lower extremity.

Ages: 19 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-02-13 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Q angle evaluation | 5 minutes
  The Q angle was measured with a standard universal goniometer. It was measured by drawing a line from the Anterior Superior Iliac Spine to the center of the patella and a second line from the center of the tibial tubercle to the center of the patella.
Electromyographic (EMG) measurements | 15 minutes
  EMG biofeedback is a device that detects neuromuscular contractions and provides feedback signals to the subject. During the ProKin 252 Techno Body balance system, Vastus Medialis and Vastus Lateralis muscles activity levels were recorded at 1000-Hz sample data-regulating Surface EMG device and analyzed using the Biometrics Datalog (UK) system.
Dynamic Balance Evaluation | 15 minutes
  Dynamic balance was evaluated by ProKin 252 Techno Body balance device. The participants were taken to the balance platform on the right foot with their eyes open, after determining the reference interval and setting the test time as 30 seconds.They were instructed to stay balanced on the platform

SECONDARY OUTCOMES:
Static Balance Evaluation | 5 minutes
  Static balance was assessed with Flamingo Balance Test (FBT) in open and closed eyes conditions.The subjects stood on the beam which was 50 cm long, 5 cm in height and 3 cm wide. Then the instructor started the stopwatch and the subjects tried to stand in this position for one minute. When the time was over, the subjects' attempts after they fell were counted and this score was recorded
Functionality Assessment | 5 minutes
  The functional status of subjects was evaluated with the Short Musculoskeletal Function Assessment Questionnaire (SMFA).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I will publish my manuscript about this study, so researchers can access my individual participant's daha with this way.

REFERENCES:
- [Background] Nguyen AD, Boling MC, Levine B, Shultz SJ. Relationships between lower extremity alignment and the quadriceps angle. Clin J Sport Med. 2009 May;19(3):201-6. doi: 10.1097/JSM.0b013e3181a38fb1. PMID 19423972